CLINICAL TRIAL: NCT06683183
Title: Ability of the Polar Wearables to Detect Fetal Heart Rate - Pilot Clinical Study
Status: Completed | Type: Observational
Sponsor: Anna Axelin (Other)
Collaborators: Polar Electro Oy (Unknown)
Responsible Party: Sponsor-Investigator, Anna Axelin, Professor, University of Turku
Organization: University of Turku (Other)
Other Study IDs: VARHA/12937/13.02.02/2024
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-11

CONDITIONS: Fetal Heart Rate Tracing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women will wear the set of wearables (chest band, smart watch and arm band) for 15 minutes. In addition, pregnant woman's ECG and fetal heart rate will be measured with hospital's patient monitor.

SUMMARY:
The aim of this clinical pilot study is

1. to evaluate the ability of the wearables to detect fetal heart rate
2. to evaluate the ability to distinguish the fetal ECG from the ECG of the mother

The participating pregnant women will wear the Polar wearables (chest band, smart watch, arm band) for 15 minutes during of which, the data will be collected with all three wearables and patient monitor (reference device). The data from the wearables will be compared with the patient monitor data referred as golden standard. Background information will be collected with questionnaires from the participants. The data collection will be conducted in hospital environment.

ELIGIBILITY:
Inclusion Criteria:

* duration of pregnancy at least 29+0 weeks
* single pregnancy
* age at least 18 years
* ability to participate in Finnish. No exclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women recruited for the study are registered at the hospital ward for pregnant women. The data collection will be conducted after the routine fetal monitoring and will not affect normal monitoring practices.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Fetal heart rate | 15 minute data collection

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided